CLINICAL TRIAL: NCT04763447
Title: Impact of Omalizumab Withdrawal After a 3 Year Duration Treatment in Well Controlled Severe Allergic Asthma : a Multicentric Randomized Controlled Trial
Brief Title: Short Treatment with Omalizumab for Severe Asthma
Acronym: SHORTEN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180614; 2024-513427-17-00 (EU CTIS Number); 2020-000883-42 (EudraCT Number)
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Asthma
Keywords: severe asthma; omalizumab; allergy; biologic
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OMA withdrawal attempt (Experimental): Patients will be told to stop abruptly (no progressive decrease of the dose) their Omalizumab treatment and they will not be prescribed new OMA
  Interventions: Other: Attempt to withdrawal OMA treatment
- OMA continuation (Active Comparator): Patients will be prescribed the same dosage of Omalizumab than they received before randomization
  Interventions: Drug: Continuation of OMA treatment

INTERVENTIONS:
Other: Attempt to withdrawal OMA treatment — Patients will be told to stop abruptly (no progressive decrease of the dose) their Omalizumab treatment and they will not be prescribed new OMA. In case of loss of control, pulmonologist can adapt asthma treatment, as in usual care. In that case, OMA can be prescribed for a second line
  Arms: OMA withdrawal attempt
Drug: Continuation of OMA treatment — Patients will be prescribed the same dosage of Omalizumab than they received before randomization, according to their weight and total circulating IgE levels.
  In case of safety concerns or loss of control, pulmonologist can modify the patient treatment regimen of OMA or other co-medications, as in usual care.
  Arms: OMA continuation

SUMMARY:
The optimal duration of the treatment by OMA remains unclear when asthma is well controlled. Data suggest that a large part of patients with well controlled asthma can discontinue OMA therapy without any asthma control deterioration or with an acceptable decrease in asthma control, therefore French experts propose that omalizumab can be given for "3 to 5 yrs if asthma remains well controlled".

The costs related to OMA are high and frequent injections represent severe constraints for patients. For all these reasons, evaluating whether shortening duration of OMA therapy is feasible while maintaining acceptable asthma control is a critical point. Therefore, the aim of this study is to evaluate asthma control after OMA discontinuation after at least 33 months of treatment when asthma is well controlled.

DETAILED DESCRIPTION:
Omalizumab (OMA) is a monoclonal anti IgE antibody, developed for severe uncontrolled allergic asthma. Efficacy of OMA in this indication is well documented in randomized trials as well as in real life studies, reducing the number of severe exacerbations by about 50% and improving asthma control score .

However, despite commercialized since 2006 in France, the optimal duration of the treatment remains unclear when asthma is well controlled. In particular, there is no guideline to apply the "step down theory" to biologics in well controlled patients.

It seems clear that a treatment given for less than one year is associated with an early relapse of the disease. However, in a randomized controlled study including 176 patients, stopping the treatment after 5 years induced a small, but acceptable loss of control (average decrease of asthma control test (ACT) by 2.88 and 1.16 point, p= 0.18), but some patients had uncontrolled asthma when the treatment was stopped. In a smaller cohort of 49 patients in Spain who voluntarily accepted to discontinue OMA treatment after 6 years of therapy, asthma deterioration (defined by one or more exacerbation and any Asthma Control Test change during the 1st year) was observed in 24% of patients during the first year following discontinuation , with a maximal rate of 2 exacerbations/yr. After 4 years of discontinuation, 60% of patients still take advantage of the 6 yrs of treatment with OMA. A retrospective study in France found that 14/26 patients treated for at least 3 years kept the same level of control after discontinuation. All these data suggest that a large part of patients with well controlled asthma can discontinue OMA therapy without any asthma control deterioration or with an acceptable decrease in asthma control.

Inducing long term asthma remissions, rather than complete cure, is one potential goal of biologics. OMA is supposed to have disease modifying effects , explaining why there is a hope for a good asthma control being maintained after discontinuation. For this reason, French experts propose that omalizumab can be given for "3 to 5 yrs if asthma remains well controlled" . After an asthma relapse, OMA can be prescribed again theoretically, but no data regarding clinical response after a "second line" of treatment with the same biologic are available. The question of optimal treatment duration is also questioned with other biologics.

The costs related to OMA are high (estimated to 12 k€/year/patient). Frequent injections (1 subcutaneous injection every 4 weeks for the lowest dose to 4 injections every 2 weeks for the highest dose) represent severe constraints for patients, especially for the youngest ones. For all these reasons, evaluating whether shortening duration of OMA therapy is feasible while maintaining acceptable asthma control is a critical point. The main objective is to demonstrate the non-inferiority (i.e. no more exacerbations at 12 months) of OMA withdrawal attempt compared to OMA continuation in asthma-controlled patients treated for at least 33 months with OMA. Secondary objectives are to compare OMA withdrawal attempt versus OMA continuation in asthma-controlled patients treated for at least 33 months with OMA on other asthma control features at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient >18 years old
* Treated with OMA, prescribed by a pulmonologist , for at least 33 months for severe allergic asthma
* Well controlled with the treatment (ACT score ⩾ 18) and having experienced no more than one exacerbation in the year preceding inclusion. An exacerbation is defined as an oral or injectable steroid course for at least 2 days and/or a minimum doubling of the usual steroid dose for at least 2 days for steroid dependent patients

Exclusion Criteria:

* Patient refusing to stop OMA treatment, whatever the reason
* Patient with other reason other than good asthma control to stop OMA, such as a side effect, planned or ongoing pregnancy, or planned switch to another step 5 asthma treatment (mepolizumab, benralizumab, dupilumab, reslizumab, daily oral steroids, bronchial thermoplasty, …)
* Patient not covered by Health Insurance
* Patient under curatorship, guardianship or safeguarding of justice
* Patient whose adherence to asthma treatments is considered poor or questionable by the investigator
* Patient participating in another intervention research
* Pregnant or lactating patient
* Patient refusing to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbations | 12 months
  Number of asthma exacerbations in the year following randomization. An exacerbation is defined as an oral or injectable steroid course for at least 2 days and/or a minimum doubling of the usual steroid dose for at least 2 days for steroid dependent patients.
  They will be assessed every 6 months from patients log book, written reports of ER visits or hospitalizations, and prescriptions

SECONDARY OUTCOMES:
Time to exacerbation | 12 months
  Number of days between the randomization and the first occurence of an exacerbation. An exacerbation is defined as an oral or injectable steroid course for at least 2 days and/or a minimum doubling of the usual steroid dose for at least 2 days for steroid dependent patients.
Asthma control (ACT) | 6 months
  Changes in asthma control test (ACT). ACT is a five questions self-administered standardized questionnaire. The ACT contains 5 questions that are related to the frequency of both asthma symptoms and required rescue medication use during the previous 4 weeks. The scores in the ACT range from 5 (worse control) to 25 (total control). A minimal change in 5 points for the total score is considered clinically significant.
Asthma control (ACT) | 12 months
  Changes in asthma control test (ACT). ACT is a five questions self-administered standardized questionnaire. The ACT contains 5 questions that are related to the frequency of both asthma symptoms and required rescue medication use during the previous 4 weeks. The scores in the ACT range from 5 (worse control) to 25 (total control). A minimal change in 5 points for the total score is considered clinically significant.
5 points-decrease of asthma control (ACT) | 6 months
  Percentage of patients with a 5 points decrease of asthma control test (ACT) compared to baseline. ACT is a five questions self-administered standardized questionnaire. The ACT contains 5 questions that are related to the frequency of both asthma symptoms and required rescue medication use during the previous 4 weeks. The scores in the ACT range from 5 (worse control) to 25 (total control). A minimal change in 5 points for the total score is considered clinically significant.
5 points-decrease of asthma control (ACT) | 12 months
  Percentage of patients with a 5 points decrease of asthma control test (ACT) compared to baseline. ACT is a five questions self-administered standardized questionnaire. The ACT contains 5 questions that are related to the frequency of both asthma symptoms and required rescue medication use during the previous 4 weeks. The scores in the ACT range from 5 (worse control) to 25 (total control). A minimal change in 5 points for the total score is considered clinically significant.
Time to loss of asthma control | 12 months
  Number of days between the randomization and the prescription of OMA (in the withdrawal group) or another step 5 asthma treatment (mepolizumab, benralizumab, daily oral steroids, bronchial thermoplasty); according to the pulmonologist's choice.
Asthma quality of life (AQLQ) | 6 months
  Changes in asthma quality of life (AQLQ). The AQLQ is a 32-item disease-specific questionnaire that has been designed to measure the functional impairments that are most troublesome to adults with asthma. Patients are asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale. The overall AQLQ score is the mean response to all 32 questions. Four independent studies have established that the AQLQ has strong measurement properties and validity.
Asthma quality of life (AQLQ) | 12 months
  Changes in asthma quality of life (AQLQ). The AQLQ is a 32-item disease-specific questionnaire that has been designed to measure the functional impairments that are most troublesome to adults with asthma. Patients are asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale. The overall AQLQ score is the mean response to all 32 questions. Four independent studies have established that the AQLQ has strong measurement properties and validity.
Number of asthma controller drugs | 6 months
  Changes in the number of asthma controller drugs
Number of asthma controller drugs | 12 months
  Changes in the number of asthma controller drugs
Dose of inhaled steroids | 6 months
  Changes in the mean daily dose of inhaled steroids received in the 3 previous months
Dose of inhaled steroids | 12 months
  Changes in the mean daily dose of inhaled steroids received in the 3 previous
Dose of oral steroids | 6 months
  Changes in the mean daily dose of oral steroids (for steroid dependent patients)
Dose of oral steroids | 12 months
  Changes in the mean daily dose of oral steroids (for steroid dependent patients)
Patients increasing their dose of oral steroids of 20% | 6 months
  Percentage of patients with a 20% increasing of the dose compared to baseline (for steroid dependent patients)
Patients increasing their dose of oral steroids of 20% | 12 months
  Percentage of patients with a 20% increasing of the dose compared to baseline (for steroid dependent patients)
Patients increasing their dose of oral steroids of 50% | 6 months
  Percentage of patients with a 50% increasing of the dose compared to baseline (for steroid dependent patients)
Patients increasing their dose of oral steroids of 50% | 12 months
  Percentage of patients with a 50% increasing of the dose compared to baseline (for steroid dependent patients)
Patients increasing their dose of oral steroids of 80% | 6 months
  Percentage of patients with a 80% increasing of the dose compared to baseline (for steroid dependent patients)
Patients increasing their dose of oral steroids of 80% | 12 months
  Percentage of patients with a 80% increasing of the dose compared to baseline (for steroid dependent patients)
Allergy manifestations | 6 months
  Occurrence of food allergy (oral syndrome and anaphylactic reactions), conjunctivitis, rhinitis, atopic dermatitis
Allergy manifestations | 12 months
  Occurrence of food allergy (oral syndrome and anaphylactic reactions), conjunctivitis, rhinitis, atopic dermatitis
FEV1 | 6 months
  Changes in FEV1
FEV1 | 12 months
  Changes in FEV1
Effect of OMA treatment duration on asthma control | 12 months
  Effet of OMA treatment duration before randomization on ACT score. The following categories will be considered: 33-48 months / 49-63 months / more than 63 months
Effect of OMA dosage on asthma control | 12 months
  Effet of OMA dosage before randomization on ACT score. The following categories will be considered: [150-300 mg/month]; ]300-600 mg/month];]600-900 mg/month] and ]900-1200 mg/month]
Effect of eosinophils rate on asthma control | 12 months
  Effet of OMA eosinophils rate at randomization on ACT score. The following categories will be considered: <300/mm3;≥300/mm3.
Effect of OMA treatment duration on time to loss of asthma control | 12 months
  Effet of OMA treatment duration before randomization on time to loss of asthma control. Time to loss of asthma control is defined as the number of days between the randomization and the prescription of OMA (in the withdrawal group) or another step 5 asthma treatment (mepolizumab, benralizumab, daily oral steroids, bronchial thermoplasty); according to the pulmonologist's choice. The following categories will be considered: 33-48 months / 49-63 months / more than 63 months
Effect of OMA dosage on time to loss of asthma control | 12 months
  Effet of OMA dosage before randomization on time to loss of asthma control. Time to loss of asthma control is defined as the number of days between the randomization and the prescription of OMA (in the withdrawal group) or another step 5 asthma treatment (mepolizumab, benralizumab, daily oral steroids, bronchial thermoplasty); according to the pulmonologist's choice. The following categories will be considered: [150-300 mg/month]; ]300-600 mg/month];]600-900 mg/month] and ]900-1200 mg/month]
Effect of eosinophils rate on time to loss of asthma control | 12 months
  Effet of OMA eosinophils rate at randomization on time to loss of asthma control. Time to loss of asthma control is defined as the number of days between the randomization and the prescription of OMA (in the withdrawal group) or another step 5 asthma treatment (mepolizumab, benralizumab, daily oral steroids, bronchial thermoplasty); according to the pulmonologist's choice. The following categories will be considered: <300/mm3;≥300/mm3.
Effect of OMA treatment duration on exacerbations | 12 months
  Effet of OMA treatment duration before randomization on exacerbations. An exacerbation is defined as an oral or injectable steroid course for at least 2 days and/or a minimum doubling of the usual steroid dose for at least 2 days for steroid dependent patients. The following categories will be considered: 33-48 months / 49-63 months / more than 63 months
Effect of OMA dosage on exacerbations | 12 months
  Effet of OMA dosage before randomization on exacerbations.An exacerbation is defined as an oral or injectable steroid course for at least 2 days and/or a minimum doubling of the usual steroid dose for at least 2 days for steroid dependent patients. The following categories will be considered: [150-300 mg/month]; ]300-600 mg/month];]600-900 mg/month] and ]900-1200 mg/month]
Effect of eosinophils rate on exacerbations | 12 months
  Effet of OMA eosinophils rate at randomization on exacerbations. An exacerbation is defined as an oral or injectable steroid course for at least 2 days and/or a minimum doubling of the usual steroid dose for at least 2 days for steroid dependent patients.The following categories will be considered: <300/mm3;≥300/mm3.
Hospitalisation for asthma | 12 months
  Number of hospitalisations for asthma in the year following randomization.
Emergency room visits for asthma | 12 months
  Emergency room visits for asthma in the year following randomization.
St. George's Respiratory Questionnaire (SGRQ) | 6 months
  Changes in St. George's Respiratory Questionnaire (SGRQ). The SGRQ is self-administered and includes 50 items in three components: symptoms, activity, and impact on daily life. The SGRQ scores range from 0 to 100, with 0 indicating no impairment in the quality of life. Higher scores on the SGRQ indicating the worst quality of life. In cohort studies, a change of four points in the total score is considered clinically significant. Many studies have established that the SGRQ is a relevant, comprehensive and content-valid instrument to assess health status in patients with severe asthma.
St. George's Respiratory Questionnaire (SGRQ) | 12 months
  Changes in St. George's Respiratory Questionnaire (SGRQ). The SGRQ is self-administered and includes 50 items in three components: symptoms, activity, and impact on daily life. The SGRQ scores range from 0 to 100, with 0 indicating no impairment in the quality of life. Higher scores on the SGRQ indicating the worst quality of life. In cohort studies, a change of four points in the total score is considered clinically significant. Many studies have established that the SGRQ is a relevant, comprehensive and content-valid instrument to assess health status in patients with severe asthma

CONTACTS AND LOCATIONS:
Overall Officials: Camille TAILLE, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal